CLINICAL TRIAL: NCT05150197
Title: Virtual Reality Visual Field Testing as an Alternative to Standard Automated Perimetry in Childhood Eye Disease
Brief Title: Virtual Reality Visual Field Testing as an Alternative in Childhood Eye Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00109426
Record Dates: First submitted 2021-11-17; First posted 2021-12-09 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Visual Field Defect, Peripheral
Keywords: Virtual Reality Visual Field; Glaucoma; Neuro-ophthalmology
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Patient (pathology) group (Experimental): This group will perform both the standard of care Humphrey Visual Field (HVF) and the VisuALL Virtual Reality Visual Field.
  Interventions: Device: VisuALL; Device: Humphrey Visual Field
- Control group (Other): This group will only perform the VisuALL Virtual Reality Visual Field.
  Interventions: Device: VisuALL

INTERVENTIONS:
Device: VisuALL — Virtual Reality Visual Field Device
Device: Humphrey Visual Field — Standard of care Visual Field test
  Arms: Patient (pathology) group

SUMMARY:
The purpose of this study is to test a new way of measuring the peripheral vision (called a visual field test) using a device which can be worn as goggles rather than being a large instrument the patient must sit at. This new visual field test (called VisuALL) is an FDA-approved virtual reality system which has been used in adults and children. This study will compare the performance of the VisuALL to the standard testing for peripheral vision, which is called the Humphrey Visual Field (HVF) test.

The study will recruit both healthy children, as well children and young adults who have eye conditions which require visual field testing as part of their standard care. The test will be performed on a day when the child or young adult already has a scheduled eye appointment as standard care. The test does not touch the eyes or require any eye drops to be given, and there is no known risk associated with the test itself. There may be a risk of loss of confidentiality. Participating in this study will require approximately 30 minutes, has no extra cost associated with it, and will be compensated by a parking pass for the day of the visit. There are no direct benefits for participants.

Selected participants will be also be given training and then loaned a home VisuALL system to allow home visual field testing. If your child is selected, additional information would be provided.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be at least four (4) years old
* Cognitively normal (no developmental delay or syndrome)
* Be able to tolerate wearing the virtual reality goggles for at least 10 minutes
* Be able to provide informed consent of a parent/guardian (and assent if 12 years or older)
* Do not have any ocular diseases that could interfere with the visual field testing

Exclusion Criteria:

* Developmental delay
* Inability to obtain consent
* Inability to understand English

Min Age: 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2022-01-19 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Mean deviation results of visual field parameters | During office visit, approximately 30 minutes
  Mean deviation of the visual field is one score measured in decibels calculated from device reading
Pattern standard deviation results of visual field parameters | During office visit, approximately 30 minutes
  Pattern standard deviation of the visual field is one score calculated from device reading
Sensitivity results of visual field parameters | During office visit, approximately 30 minutes
  Sensitivities are the results of each space in the visual field measured in decibels

SECONDARY OUTCOMES:
Percent of times that scotomas were visualized as measured by visual field tests | During office visit, approximately 30 minutes
Percent of participants stating satisfaction as measured by questionnaire | During office visit, approximately 5 minutes
  12 questions with strongly disagree to strongly agree
Percent of patients able to use VisuALL home testing as measured by device reading | One month, 1-2 tests per week
  Home testing will be done in a few patients that demonstrate facility with device
Percent of patients able to use VisuALL in-office testing as measured by patient observation | During office visit, approximately 30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Sharon F Freedman, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Razeghinejad R, Gonzalez-Garcia A, Myers JS, Katz LJ. Preliminary Report on a Novel Virtual Reality Perimeter Compared With Standard Automated Perimetry. J Glaucoma. 2021 Jan 1;30(1):17-23. doi: 10.1097/IJG.0000000000001670. PMID 32941320
- [Background] Montelongo M, Gonzalez A, Morgenstern F, Donahue SP, Groth SL. A Virtual Reality-Based Automated Perimeter, Device, and Pilot Study. Transl Vis Sci Technol. 2021 Mar 1;10(3):20. doi: 10.1167/tvst.10.3.20. PMID 34003954